CLINICAL TRIAL: NCT04784091
Title: Randomized, Controlled, Multicenter, Double-Masked, Parallel, Phase 3 Trial to Evaluate the Safety and Efficacy of TP-03 for the Treatment of Demodex Blepharitis
Brief Title: Trial to Evaluate the Safety and Efficacy of TP-03 for the Treatment of Demodex Blepharitis
Acronym: Saturn-2
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Tarsus Pharmaceuticals, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: TRS-010
Record Dates: First submitted 2021-03-02; First posted 2021-03-05 (Actual); Results first posted 2023-12-21 (Actual); Last update posted 2023-12-21 (Actual); Status verified 2023-12

CONDITIONS: Blepharitis
Keywords: Demodex
MeSH Terms: conditions — Blepharitis

STUDY DESIGN:
Intervention Model Description: Active arm: TP-03, 0.25% Control arm: Vehicle of TP-03
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: Treatment assignment will be unknown to the study participant, investigators and site staff performing study assessments.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Active (Experimental): TP-03, lotilaner ophthalmic solution, 0.25%, administered topically twice a day for approximately 43 days
  Interventions: Drug: TP-03
- Control (Placebo Comparator): Vehicle of TP-03 ophthalmic solution, administered topically twice a day for approximately 43 days
  Interventions: Drug: TP-03 Vehicle

INTERVENTIONS:
Drug: TP-03 — TP-03, lotilaner ophthalmic solution, 0.25%, administered twice a day
  Arms: Active
Drug: TP-03 Vehicle — Vehicle of TP-03 ophthalmic solution, administered twice a day
  Arms: Control

SUMMARY:
The purpose of this study is to compare the safety and efficacy of TP-03, an eyedrop, to its vehicle control for the treatment of blepharitis due to Demodex, a microscopic mite frequently found in human hair follicles.

DETAILED DESCRIPTION:
This Phase 3 study is a randomized, controlled, multicenter, double-masked, parallel trial to compare the safety and efficacy of TP-03 to vehicle control for the treatment of Demodex blepharitis. The primary objective of the study is to assess the safety and efficacy of TP-03, 0.25% compared to its vehicle from Day 1 to Day 43 in adult participants with mild to severe Demodex blepharitis. The primary efficacy endpoint will be cure based upon collarettes. Safety will be determined by assessing adverse effects related to the treatment as well as evaluating any changes in visual acuity, intraocular pressure, slit lamp biomicroscopy, endothelial cell density, hematology, blood chemistry, and urinalysis.

ELIGIBILITY:
Inclusion Criteria:

* Be willing to sign the informed consent and deemed capable of complying with the requirements of the study protocol
* Meet all of the following criteria in at least one eye: Have more than 10 lashes with collarettes present on the upper lid; have at least mild erythema of the upper eyelid margin; have an average Demodex density, upper and lower eyelids combined, of 1.5 or more mites per lash

Exclusion Criteria:

* Have used lid hygiene products within 14 days of Screening or unwilling to forego the use of lid hygiene products during the study
* Have used a prostaglandin analogue to promote eyelash growth within 30 days of Screening or any plans to initiate treatment during the study
* Have used artificial eyelashes or eyelash extensions within 7 days of Screening or be unwilling to forego their use during the study
* Be pregnant or lactating at the time of Screening

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 412 (Actual)
Dates: Start 2021-04-29 (Actual); Primary Completion 2022-05-09 (Actual); Study Completion 2022-05-09 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: John Meyer, MD, Principal Investigator — The Eye Care Institute
Locations (21):
- United States (21):
  - Global Retina Institute, Scottsdale, Arizona
  - Shultz Chang Vision, Northridge, California
  - East Bay Eye Center, San Ramon, California
  - Vision Institute, Colorado Springs, Colorado
  - Pinnacle Research Institute, Fort Lauderdale, Florida
  - Jackson Eye, S.C., Lake Villa, Illinois
  - Pankratz Eye Institute, Columbus, Indiana
  - Michael Washburn Center for Ophthalmic Research LLC, Indianapolis, Indiana
  - Kannarr Eye Care, Pittsburg, Kansas
  - The Eye Care Institute, Louisville, Kentucky
  - Complete Eye Care of Medina, Medina, Minnesota
  - Tauber Eye Center, Kansas City, Missouri
  - Ophthalmology Associates, St Louis, Missouri
  - NC Eye Associates, Apex, North Carolina
  - Pure Ophthalmic Research, Mint Hill, North Carolina
  - Vita Eye Clinic, Shelby, North Carolina
  - Northern Ophthalmic Associates, Jenkintown, Pennsylvania
  - Alpine Research Organization / Healthy Heart Clinics of America, Clinton, Utah
  - Alpine Research Organization Inc./ Country Hills Eye Center, Ogden, Utah
  - Periman Eye Institute, Seattle, Washington
  - New River Vision Care, Oak Hill, West Virginia

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Gaddie IB, Donnenfeld ED, Karpecki P, Vollmer P, Berdy GJ, Peterson JD, Simmons B, Edell ARP, Whitson WE, Ciolino JB, Baba SN, Holdbrook M, Trevejo J, Meyer J, Yeu E; Saturn-2 Study Group. Lotilaner Ophthalmic Solution 0.25% for Demodex Blepharitis: Randomized, Vehicle-Controlled, Multicenter, Phase 3 Trial (Saturn-2). Ophthalmology. 2023 Oct;130(10):1015-1023. doi: 10.1016/j.ophtha.2023.05.030. Epub 2023 Jun 5. PMID 37285925

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Active | Control
Started | 203 | 209
Completed | 193 | 200
Not Completed | 10 | 9

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Active | Control | Total
Number analyzed (Participants) | 203 | 209 | 412
Age, Continuous [Mean (Standard Deviation); unit: years] | 63.9 (15.15) | 65.1 (13.35) | 64.5 (14.26)
Age, Customized [Count of Participants; unit: Participants]
  < 65 years | 84 | 80 | 164
  ≥ 65 years | 119 | 129 | 248
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 97 | 103 | 200
  Male | 106 | 106 | 212
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 17 | 17 | 34
  Not Hispanic or Latino | 186 | 192 | 378
  Unknown or Not Reported | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 1 | 1 | 2
  Asian | 3 | 3 | 6
  Native Hawaiian or Other Pacific Islander | 2 | 0 | 2
  Black or African American | 20 | 15 | 35
  White | 176 | 187 | 363
  More than one race | 1 | 0 | 1
  Unknown or Not Reported | 0 | 3 | 3
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 203 | 209 | 412

OUTCOME MEASURES:

1. Primary Outcome: The Proportion of Participants Cured Based on Their Collarette Score of 0 for the Upper Eyelid.
Description: The proportion of subjects cured where cure is defined as 0-2 lashes with collarettes on the upper eyelid of the analysis eye.
  The primary outcome analysis is the combined result from 20 analyses each with missing data imputed. Missing data were imputed per the method described in the SAP. The least square mean is computed from the result of the 20 analyses with imputed missing values
Time Frame: 43 days
Measure: Least Squares Mean (Standard Error); unit: Proportion cured
Arm/Group | Active | Control
Number analyzed (Participants) | 203 | 209
Proportion cured | 0.547 (0.035) | 0.122 (0.023)

2. Secondary Outcome: The Proportion of Participants With Their Demodex Mites Eradicated.
Description: The proportion of participants with Demodex mites eradicated at Day 43 where eradication is defined as a mite density of 0 mites/lash for the analysis eye. The mite density is obtained by epilating four of more lashes and dividing the number of mites observed under the microscope by the number of lashes.
  The primary outcome analysis is the combined result from 20 analyses each with missing data imputed. Missing data were imputed per the method described in the SAP. The least square mean is computed from the result of the 20 analyses with imputed missing values
Time Frame: 43 days
Measure: Least Squares Mean (Standard Error); unit: Proportion eradicated
Arm/Group | Active | Control
Number analyzed (Participants) | 203 | 209
Proportion eradicated | 0.499 (0.036) | 0.14 (0.024)

3. Secondary Outcome: The Proportion of Participants Cured Based on a Composite of Collarette Score and Erythema Score
Description: The proportion of participants cured where cure is defined as a composite of the collarettes, 0-2 lashes with collarettes on the upper eyelid of the analysis eye, and normal lid margin erythema for the upper eyelid of the analysis eye at Day 43.
  The primary outcome analysis is the combined result from 20 analyses each with missing data imputed. Missing data were imputed per the method described in the SAP. The least square mean is computed from the result of the 20 analyses with imputed missing values.
Time Frame: 43 days
Measure: Median (Standard Error); unit: Proportion cured
Arm/Group | Active | Control
Number analyzed (Participants) | 203 | 209
Proportion cured | 0.187 (0.028) | 0.039 (0.014)

4. Secondary Outcome: The Proportion of Participants Cured Based on Erythema Score.
Description: The proportion of participants cured based on erythema where cure is defined as having a normal eyelid erythema of the analysis eye at day 43.
  The primary outcome analysis is the combined result from 20 analyses each with missing data imputed. Missing data were imputed per the method described in the SAP. The least square mean is computed from the result of the 20 analyses with imputed missing values.
Time Frame: 43 days
Measure: Least Squares Mean (Standard Error); unit: Proportion cured
Arm/Group | Active | Control
Number analyzed (Participants) | 203 | 209
Proportion cured | 0.303 (0.033) | 0.091 (0.02)

ADVERSE EVENTS:
Time Frame: 90 Days
Arm/Group | Active | Control
All-Cause Mortality (participants affected / at risk) | 0/203 | 0/209
Serious Adverse Events (participants affected / at risk) | 4/203 | 3/209
Other Adverse Events (participants affected / at risk) | 49/203 | 28/209
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Active (N=203) | Control (N=209)
Diabetic retinopathy (Eye disorders) | 1 | 0
Gastrointestinal haemorrhage (Gastrointestinal disorders) | 1 | 0
Bladder Cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Uterine prolapse (Reproductive system and breast disorders) | 1 | 0
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Intestinal obstruction (Gastrointestinal disorders) | 1 | 0
Covid-19 (Infections and infestations) | 0 | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 1% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Active (N=203) | Control (N=209)
Visual acuity reduced (Eye disorders) | 5 | 6
Dry eye (Eye disorders) | 4 | 2
Punctate keratitis (Eye disorders) | 4 | 1
Chalazion (Eye disorders) | 3 | 0
Conjunctival haemorrhage (Eye disorders) | 2 | 1
Conjunctival hyperaemia (Eye disorders) | 3 | 0
Eyelid oedema (Eye disorders) | 3 | 1
Instillation site pain (General disorders) | 16 | 13
Hordeolum (Infections and infestations) | 4 | 1
Seasonal allergy (Immune system disorders) | 2 | 1
Urinary tract infection (Infections and infestations) | 3 | 2
Nasopharyngitis (Infections and infestations) | 3 | 1
SARS-CoV-2 test positive (Investigations) | 3 | 1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
It is specified in the protocol that the data generated in this clinical trial, all related information and any materials containing such data and information are the exclusive property of Tarsus Pharmaceuticals, Inc. and are confidential to Tarsus Pharmaceuticals. Also, the investigator or other study-related personnel may not disclose to anyone or use any data, information or materials related to this clinical trial without the express written consent of Tarsus Pharmaceuticals.

DOCUMENTS (2):
  • Study Protocol (2021-12-09): https://cdn.clinicaltrials.gov/large-docs/91/NCT04784091/Prot_003.pdf
  • Statistical Analysis Plan (2022-03-22): https://cdn.clinicaltrials.gov/large-docs/91/NCT04784091/SAP_004.pdf